CLINICAL TRIAL: NCT01880567
Title: A Phase II Study of Ibrutinib Plus Rituximab in Patients With Relapsed/Refractory Mantle Cell Lymphoma or Elderly Patients With Newly Diagnosed MCL
Brief Title: Ibrutinib and Rituximab in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma or Older Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0090; NCI-2013-01304 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0090 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: CCND1 Positive; CCND2 Positive; CCND3 Positive; CD20 Positive; Mantle Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, rituximab) (Experimental): Patients receive ibrutinib PO daily on days 1-28 and rituximab IV over 4-8 hours on days 1, 8, 15, and 22 of course 1; on day 1 of courses 3-8; and on day 1 of every other course for all subsequent courses. Treatment with rituximab repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Courses with ibrutinib repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies how well ibrutinib and rituximab work in treating patients with mantle cell lymphoma that has come back or has not responded to treatment or older patients with newly diagnosed mantle cell lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, may find cancer cells and help kill them. Giving ibrutinib and rituximab may be an effective treatment for mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate of ibrutinib plus rituximab in patients with relapsed and/or refractory mantle cell lymphoma (MCL).

II. To evaluate the safety and response rate of ibrutinib plus rituximab in elderly patients (> 65) with newly-diagnosed, untreated MCL.

SECONDARY OBJECTIVES:

I. To further evaluate the toxicity profile of the combination of ibrutinib and rituximab in patients with relapsed and/or refractory MCL.

II. To estimate the overall response rate (ORR); (partial response [PR] or better), the response duration (DOR), progression-free survival (PFS), time to progression (TTP) and overall survival (OS) in patients with relapsed and/or refractory MCL; clinical benefit response (CBR) = (minimal response [MR] + ORR) will also be evaluated.

III. To estimate the response duration, PFS, time to progression (TTP), and OS in elderly patients (> 65) with newly-diagnosed, untreated MCL.

EXPLORATORY OBJECTIVES:

I. To correlate detected gene mutations and changes in gene and/or protein expression with response to treatment.

OUTLINE:

Patients receive ibrutinib orally (PO) daily on days 1-28 and rituximab intravenously (IV) over 4-8 hours on days 1, 8, 15, and 22 of course 1; on day 1 of courses 3-8; and on day 1 of every other course for all subsequent courses. Treatment with rituximab repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Courses with ibrutinib repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory MCL: Confirmed diagnosis of mantle cell lymphoma with cluster of differentiation (CD)20 and cyclin D1 through cyclin D3 positivity in tissue biopsy
* Relapsed/refractory MCL: Patient has relapsed and or refractory MCL and must have received at least one prior treatment regimen for their disease; patient with leukemia phase (peripheral blood involvement), leptomeningeal disease, cerebral spinal fluid (CSF) MCL, central nervous system (CNS) MCL, non-measurable disease, gastrointestinal (GI) MCL, or bone marrow (BM) MCL are also eligible
* Relapsed/refractory MCL: Understand and voluntarily sign an Institutional Review Board (IRB)-approved informed consent form
* Relapsed/refractory MCL: Patients with bone marrow or gastrointestinal (GI) only involvement are acceptable
* Relapsed/refractory MCL: Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Relapsed/refractory MCL: Absolute neutrophil count (ANC) >= 500/mm^3; (patients who have bone marrow infiltration by MCL are eligible if their ANC is >= 500/mm^3 [growth factor allowed]; these patients should be discussed with either the principal investigator [PI] or Co-PI of the study for final approval)
* Relapsed/refractory MCL: Platelet count >= 30,000/mm^3 (transfusion to reach platelet count allowed); (patients who have bone marrow infiltration by MCL are eligible if their platelet level is equal to or > than 15,000/mm^3; these patients should be discussed with either the PI or Co-PI of the study for final approval)
* Relapsed/refractory MCL: Aspartate transaminase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present
* Relapsed/refractory MCL: Serum bilirubin < 1.5 mg/dl
* Relapsed/refractory MCL: Creatinine (Cr) clearance >= 30 mL/min
* Relapsed/refractory MCL: Patients must be willing to receive transfusions of blood products
* Relapsed/refractory MCL: Willing and able to participate in all study related procedures and therapy including swallowing capsules without difficulty
* Newly diagnosed MCL: Confirmed diagnosis of MCL with CD20 and cyclin D1 positivity in tissue biopsy; patients must have never received any prior therapy for their disease
* Newly diagnosed MCL: Understand and voluntarily sign an IRB-approved informed consent form
* Newly diagnosed MCL: Age > 65 years at the time of signing the informed consent
* Newly diagnosed MCL: Patients should in general have bi-dimensional measurable disease with their biggest tumor less than 10 cm; (bone marrow or gastrointestinal [GI] only involvement is acceptable)
* Newly diagnosed MCL: Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Newly diagnosed MCL: Absolute neutrophil count (ANC) > 750/mm^3; patients who have bone marrow infiltration by MCL are eligible if their ANC is equal to or > than 500
* Newly diagnosed MCL: Platelet count > 50,000/mm^3; patients who have bone marrow infiltration by MCL are eligible if their platelet level is equal to or > than 15,000 /mm^3; (platelet transfusions are allowed; these patients should be discussed with either the PI or Co-PI of the study for final approval)
* Newly diagnosed MCL: AST (SGOT) and ALT (SGPT) < 2 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present
* Newly diagnosed MCL: Uric acid within normal limits (allopurinol is allowed to bring abnormal level to within normal limits)
* Newly diagnosed MCL: Serum bilirubin < 1.5 mg/dl
* Newly diagnosed MCL: Creatinine (Cr) Clearance >= 30 mL/min
* Newly diagnosed MCL: Ki67 protein (Ki67) < 50%
* Newly diagnosed MCL: Disease free of prior malignancies of equal to or greater than 6 months with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years
* Newly diagnosed MCL: Patients must be willing to receive transfusions of blood products
* Newly diagnosed MCL: Willing and able to participate in all study related procedures and therapy including swallowing capsules without difficulty

Exclusion Criteria:

* Relapsed/refractory MCL: Any serious medical condition that places the patient at unacceptable risk and/or would prevent the subject from signing the informed consent form; examples include but are not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, active infection, active hemorrhage, or psychiatric illness
* Relapsed/refractory MCL: Pregnant or breast feeding females
* Relapsed/refractory MCL: Known human immunodeficiency virus (HIV) infection; patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody); known hepatitis C infection is allowed as long as there is no active disease and is cleared by gastrointestinal (GI) consultation
* Relapsed/refractory MCL: The patient has a prior or concurrent malignancy that in the opinion of the investigator, presents a greater risk to the patient's health and survival, than of the MCL, within the subsequent 6 months at the time of consent
* Relapsed/refractory MCL: History of stroke or intracranial hemorrhage within 6 months prior to signing the consent
* Relapsed/refractory MCL: Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months at the time of consent or any class 3 (moderate) or 4 (severe) cardiac disease defined by the New York Heart Association classification
* Relapsed/refractory MCL: Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, bradycardia (< 50 beats per minute [bpm]), or corrected QT (QTc) > 500 msec
* Relapsed/refractory MCL: Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Relapsed/refractory MCL: Prior chemotherapy within 3 weeks, nitrosoureas within 6 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy or other investigational agents within 3 weeks, major surgery within 4 weeks or vaccination with live attenuated vaccines within 4 weeks of the first dose of study drug
* Relapsed/refractory MCL: Prior treatment with ibrutinib
* Relapsed/refractory MCL: Requires anticoagulation with warfarin or equivalent vitamin K antagonist
* Relapsed/refractory MCL: Requires treatment with strong cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) inhibitors
* Newly Diagnosed MCL: Any serious medical condition that places the patient at unacceptable risk and/or would prevent the subject from signing the informed consent form; examples include but are not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, active infection requiring treatment with systemic antibiotics, antiviral or antifungal agents, active hemorrhage, or psychiatric illness
* Newly diagnosed MCL: Known HIV infection; patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody); known hepatitis C infection is allowed as long as there is no active disease and is cleared by GI consultation
* Newly diagnosed MCL: The patient has a prior or concurrent malignancy that in the opinion of the investigator, presents a greater risk to the patient's health and survival, than of the MCL, within the subsequent 6 months at the time of consent
* Newly diagnosed MCL: History of stroke or intracranial hemorrhage within 6 months prior to signing the consent
* Newly diagnosed MCL: Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months at the time of consent or any class 3 (moderate) or 4 (severe) cardiac disease defined by the New York Heart Association Classification
* Newly diagnosed MCL: Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree AV block type II, 3rd degree block, bradycardia (< 50 bpm), or QTc > 500 msec
* Newly diagnosed MCL: Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Newly diagnosed MCL: Major surgery within 4 weeks or vaccination with live attenuated vaccines within 4 weeks of the first dose of study drug
* Newly diagnosed MCL: Prior treatment with ibrutinib
* Newly diagnosed MCL: Requires concomitant anticoagulation with warfarin or equivalent vitamin K antagonist
* Newly diagnosed MCL: Requires treatment with strong CYP3A4/5 inhibitors
* Newly diagnosed MCL: Patients with blastoid and pleomorphic variants
* Newly diagnosed MCL: Ki-67 to be equal or more than 50%
* Newly diagnosed MCL: Central nervous system lymphoma
* Newly diagnosed MCL: Patients with bi-dimensional measurable disease with a tumor >= 10 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall response (complete response and partial response), assessed by the International Workshop Standardized Response Criteria for non-Hodgkin lymphoma | Up to 8 weeks
  Overall response will be monitored using the Bayesian stopping boundaries calculated based on beta-binomial distribution.
Overall response (complete response and partial response) in elderly patients with newly-diagnosed, untreated mantle cell lymphoma, assessed by the International Workshop Standardized Response Criteria for non-Hodgkin lymphoma | Up to 8 weeks
  Overall response will be monitored using the Bayesian stopping boundaries calculated based on beta-binomial distribution.
Incidence of toxicity, defined as grade 3 or higher non-hematologic toxicity, grade 3 neutropenia, grade 4 hematologic toxicity, inability to administer full schedule and dose, or inability to receive treatment day 1 of course 2 | Up to 4 weeks
  Toxicity data will be summarized by frequency tables for all patients.
Incidence of grade 3 or higher non-hematologic toxicity, grade 3 neutropenia, grade 4 hematologic toxicity, inability to administer full schedule and dose, or inability to receive treatment day 1 of course 2 in newly diagnosed elderly patients | Up to 4 weeks
  Toxicity data will be summarized by frequency tables for all patients.

SECONDARY OUTCOMES:
Clinical benefit response (minimal response + overall response rate), | Up to 6 years
  Will be assessed by the International Workshop Standardized Response Criteria for non-Hodgkin lymphoma.
Duration of response | Up to 6 years
  Duration of response will be estimated using the method of Kaplan and Meier. Comparison by important subgroups will be made using the log-rank test. Cox proportional hazards will be employed for multivariate analysis.
Progression-free survival | Up to 6 years
  Progression-free survival will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazard regression will be employed for multivariate analysis on time-to-events outcomes.
Time to progression | Up to 6 years
  Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazard regression will be employed for multivariate analysis on time-to-events outcomes.
Overall survival | Up to 6 years
  Overall survival will be estimated using the method of Kaplan and Meier. Comparison by important subgroups will be made using the log-rank test. Cox proportional hazards will be employed for multivariate analysis.
Duration of response in elderly patients with newly diagnosed, untreated mantle cell lymphoma | Up to 6 years
  Intend-to-treat analysis will be applied to the eligible patients.
Progression-free survival in elderly patients with newly diagnosed, untreated mantle cell lymphoma | Up to 6 years
  Intend-to-treat analysis will be applied to the eligible patients.
Overall survival in elderly patients with newly diagnosed, untreated mantle cell lymphoma | Up to 6 years
  Overall response will be monitored using the Bayesian stopping boundaries calculated based on beta-binomial distribution.
Time to progression in elderly patients with newly diagnosed, untreated mantle cell lymphoma | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Preetesh Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Zhao S, Lee HJ, Hill HA, Ok CY, Kanagal-Shamanna R, Hagemeister FB, Fowler N, Fayad L, Yao Y, Liu Y, Moghrabi OB, Navsaria L, Feng L, Nogueras Gonzalez GM, Xu G, Thirumurthi S, Santos D, Iliescu C, Tang G, Medeiros LJ, Vega F, Avellaneda M, Badillo M, Flowers CR, Wang L, Wang ML. Ibrutinib With Rituximab in First-Line Treatment of Older Patients With Mantle Cell Lymphoma. J Clin Oncol. 2022 Jan 10;40(2):202-212. doi: 10.1200/JCO.21.01797. Epub 2021 Nov 19. PMID 34797699
- [Derived] Wang ML, Lee H, Chuang H, Wagner-Bartak N, Hagemeister F, Westin J, Fayad L, Samaniego F, Turturro F, Oki Y, Chen W, Badillo M, Nomie K, DeLa Rosa M, Zhao D, Lam L, Addison A, Zhang H, Young KH, Li S, Santos D, Medeiros LJ, Champlin R, Romaguera J, Zhang L. Ibrutinib in combination with rituximab in relapsed or refractory mantle cell lymphoma: a single-centre, open-label, phase 2 trial. Lancet Oncol. 2016 Jan;17(1):48-56. doi: 10.1016/S1470-2045(15)00438-6. Epub 2015 Nov 28. PMID 26640039
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org